CLINICAL TRIAL: NCT03557749
Title: Monitoring of Immune and Microbial Reconstitution in Hematopoietic Cell Transplantation (HCT) and Novel Immunotherapies
Brief Title: Monitoring of Immune and Microbial Reconstitution in (HCT) and Novel Immunotherapies
Status: Terminated | Type: Observational
Why Stopped: Accrual goal met
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2017NTLS045; MT2017-12 (Other: Masonic Cancer Center, University of Minnesota)
Record Dates: First submitted 2018-05-15; First posted 2018-06-15 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Immune and Microbial Reconstitution; Systemic Viral Infection; Acute-graft-versus-host Disease; Chronic Graft-versus-host-disease; Recurrent Malignancy; Cytokine Release Syndrome; Allogenic Related Donors; Cell Therapy/Immunotherapy Patients
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Neoplasms; Cytokine Release Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Immune and Microbial Reconstitution
  Interventions: Diagnostic Test: Blood Sample; Diagnostic Test: Stool Sample; Diagnostic Test: Urine Sample
- Immune Response Triggered by Severe, Systemic Viral Infection
  Interventions: Diagnostic Test: Blood Sample; Diagnostic Test: Bronchoalveolar Lavage (BAL) fluid
- Immune Response Triggered by Acute Graft-versus-Host Disease
  Interventions: Diagnostic Test: Blood Sample; Diagnostic Test: Stool Sample; Diagnostic Test: Gastrointestinal biopsy x 2-4; Diagnostic Test: Skin biopsy
- Immune Response Triggered by Chronic Graft-versus-Host Disease
  Interventions: Diagnostic Test: Blood Sample; Diagnostic Test: Skin biopsy; Diagnostic Test: Skin, mouth, and/or ocular swab
- Immune Response Triggered by Relapse
  Interventions: Diagnostic Test: Blood Sample
- Immune Response Triggered by Cytokine Release Syndrome
  Interventions: Diagnostic Test: Blood Sample
- Allogeneic Related Donor Samples
  Interventions: Diagnostic Test: Blood Sample; Diagnostic Test: Stool Sample; Diagnostic Test: Urine Sample
- Cellular Therapy Products
  Interventions: Diagnostic Test: Apheresis Product; Diagnostic Test: Final cellular product

INTERVENTIONS:
Diagnostic Test: Blood Sample — 60 ml heparinized blood 10 ml serum
  Groups: Allogeneic Related Donor Samples; Immune Response Triggered by Acute Graft-versus-Host Disease; Immune Response Triggered by Chronic Graft-versus-Host Disease; Immune Response Triggered by Cytokine Release Syndrome; Immune Response Triggered by Relapse; Immune Response Triggered by Severe, Systemic Viral Infection; Immune and Microbial Reconstitution
Diagnostic Test: Stool Sample — pea-sized amount
  Groups: Allogeneic Related Donor Samples; Immune Response Triggered by Acute Graft-versus-Host Disease; Immune and Microbial Reconstitution
Diagnostic Test: Urine Sample — 10 ml
  Groups: Allogeneic Related Donor Samples; Immune and Microbial Reconstitution
Diagnostic Test: Bronchoalveolar Lavage (BAL) fluid — 10 ml
  Groups: Immune Response Triggered by Severe, Systemic Viral Infection
Diagnostic Test: Gastrointestinal biopsy x 2-4 — rectosigmoid site preferred
  Groups: Immune Response Triggered by Acute Graft-versus-Host Disease
Diagnostic Test: Skin biopsy — 2-4 mm punch
  Groups: Immune Response Triggered by Acute Graft-versus-Host Disease; Immune Response Triggered by Chronic Graft-versus-Host Disease
Diagnostic Test: Skin, mouth, and/or ocular swab — Involved skin, mouth, and/or ocular swab for microbiota studies
  Groups: Immune Response Triggered by Chronic Graft-versus-Host Disease
Diagnostic Test: Apheresis Product — Up to 10 ml of apheresis product
  Groups: Cellular Therapy Products
Diagnostic Test: Final cellular product — A second washing from the infusion bag after product and initial bag wash has infused, or up to 10 ml of final cellular product
  Groups: Cellular Therapy Products

SUMMARY:
This protocol serves as a mechanism to collect, store, and distribute bodily fluid and tissue samples obtained from Hematopoietic Cell Transplant (HCT) or novel immunotherapy patients and their donors at the Masonic Cancer Center in order to conduct correlative studies of the immune system, microbiota, and their interactions. Fluid (including but not limited to, blood, urine, saliva, cerebrospinal fluid, bronchoalveolar lavage fluid) sample log-in, processing, relabeling, and storage is performed by the Masonic Cancer Center (MCC) Translational Therapy Lab (TTL).

ELIGIBILITY:
Inclusion Criteria:

* Patients planning to undergo HCT or other cellular therapy/immunotherapy
* Allogeneic related donors
* Aged 0-80
* Willing and able to sign voluntary written consent

Exclusion Criteria:

* Patients whose medical record indicates that they have opted out of research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving care in the University of Minnesota Blood and Marrow Transplant Program
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Immune Function after HCT | 7 Years
  Incidence of neutrophil recovery
Immune Function after HCT | 7 Years
  Incidence of lymphocyte and monocyte subset recovery
Immune Function after HCT | 7 Years
  Incidence of grade II-IV acute GVHD
Immune Function after HCT | 7 Years
  Incidence of CMV reactivation
Immune Function after Cell Therapy/Immunotherapy | 7 Years
  Incidence of neutrophil recovery
Immune Function after Cell Therapy/Immunotherapy | 7 Years
  Incidence of lymphocyte and monocyte subset recovery
Immune Function after Cell Therapy/Immunotherapy | 7 Years
  Incidence of cytokine release syndrome (CRS)
Correlate Immune Parameters | 7 Years
  Correlate the lymphocyte phenotypes, specifically natural killer cell subsets and lymphocyte response to viral antigen.
Correlate microbiota changes and their interactions with the host with outcomes of HCT | 7 Years
  Correlate microbiota changes and their interactions with the host with outcomes of HCT

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States